CLINICAL TRIAL: NCT04321291
Title: Impact of a Nurse's Specific Information on the Acceptability of Biosimilars in Chronic Inflammatory Rheumatism
Brief Title: Information and Acceptability of Biosimilars
Acronym: BIOSIMINFO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RECHMPL19_0084
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Rheumatoid Arthritis; Spondyloarthritis; Psoriatic Arthritis
Keywords: Rheumatoid arthritis; Spondyloarthritis; Biologics; Biosimilars information
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylarthritis; Arthritis, Psoriatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurse information (Experimental): The patient will receive a generic information leaflet plus an Individual information by nurse on biosimilars
  Interventions: Other: Individual information by nurse on biosimilars
- Information Leaflet (Other): The patient will receive a generic information leaflet only
  Interventions: Other: Generic information leaflet

INTERVENTIONS:
Other: Generic information leaflet — The information about the biosimiliars is realized only by the transmission of the information leaflet in addition to the information given by the investigator.
  Arms: Information Leaflet
Other: Individual information by nurse on biosimilars — Delivery of the same information leaflet, completed if asked by the patient, by individual meeting with specialist nurse, including generic and standardized informations on specificities, advantages and current scientific knowledge about biosimilars in inflammatory rheumatic diseases. This is in addition to the information given by the investigator
  Arms: Nurse information

SUMMARY:
Patients with rheumatoid arthritis or spondyloarthritis, currently treated or about to be started with anti-TNF original drug adalimumab or etanercept will be included and randomized to either " information leaflet only " or " information leaflet + nurse information " arms, just before they see their rheumatologist for periodic assessment of disease and treatment.

Patients from the " information leaflet only " arm will be distributed individually a dedicated leaflet with written generic informations about the use of biosimilars in rheumatic diseases (individual and societal advantages, pharmaceutical development, scientific efficacy and safety results).

Patients from the " " information leaflet + nurse information " arm will be delivered the same leaflet, and additionally offered to have a dedicated individual interview with a specialist nurse, who will orally discuss informations about biosimilars based on a standardized talk, completed by answers to any questions by the patient.

The rheumatologist will then propose, unless inappropriate based on clinical evaluation of the patient, a change in the treatment of patients from the original drug to the corresponding biosimilar.

The primary outcome will be the observed proportions of patients actually receiving the biosimilar drug at the 6-months follow-up visit in the 2 compared arms.

Secondary outcomes will be average time spent by the nurse to adequatley inform the patient, the proportion of patients from the intervention arm who have actually asked for the nurse information interview, and the reasons for refusal of biosimilars, when appropriate.

ELIGIBILITY:
Inclusion criteria:

* Age 18 and over (no upper age limit)
* All adult patients seen in rheumatology consultation at the Montpellier Hospital
* With inflammatory rheumatism (rheumatoid arthritis or spondyloarthritis).
* Treated (or in the process of being treated at the end of the consultation) by etanercept or adalimumab
* In whom the biomedical treatment already used should in principle be renewed without modification (patient deemed good responder and well tolerant of the treatment)
* Or where biomedical initiation has just been indicated during the consultation
* Member of a social security scheme
* Informed and written consent

Exclusion criteria:

* Unable to understand information (not fluent in the French language, severe cognitive impairment, etc.)
* Known intolerance to one of the proposed biosimilar excipients
* Vulnerable persons: pregnant woman, minor patient, deprived of liberty, under guardianship or under curatorship

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2020-07-02 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Observed rate of prescribed biosimilars | 18 months
  The measure is the number of patient who accept the biosimilars

SECONDARY OUTCOMES:
Average time spent by nurse to inform patients | 18 months
  the measure is done by the completion of a questionnaire by the nurse who report the time spent with the patient
Proportion of patients from the intervention arm having actually received specific information by nurse | 18 months
  Verify the number of patient who receive the information thanks to the nurse questionnaire
Reasons for refusal of biosimilars | 18 months
  The measure is done by the completion of a questionnaire by the patient

CONTACTS AND LOCATIONS:
Overall Officials: Cédric LUKAS, Principal Investigator — Montpellier University Hospital
Locations (1):
- CHU, Service Immuno-rhumatologie, Département de rhumatologie, Montpellier, France

IPD SHARING:
Plan to Share IPD: No